CLINICAL TRIAL: NCT05737199
Title: A Single-arm Open-label Phase II Trial to Assess the Efficacy and Safety of Pembrolizumab for Unresectable Advanced or Recurrent Ovarian Squamous Cell Carcinoma
Brief Title: Assessment of the Efficacy and Safety of Pembrolizumab for Ovarian Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Niigata University Medical & Dental Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Kosuke Yoshihara, Professor, Niigata University Medical & Dental Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JGOG3029
Record Dates: First submitted 2023-02-12; First posted 2023-02-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Squamous Cell Carcinoma
Keywords: Pembrolizumab
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MK-3475 (Pembrolizumab) (Experimental): Treatment with MK-3475 (pembrolizumab) 200 mg.
  Interventions: Drug: MK-3475 (pembrolizumab)

INTERVENTIONS:
Drug: MK-3475 (pembrolizumab) — MK-3475 (pembrolizumab) 200mg IV every 3 weeks [Q3W] Treated for 2 years (35 cycles), or until PD, unacceptable toxicity, or study withdrawal.
  Other Names: Keytruda

SUMMARY:
This is a phase II, non-randomized, open-label, single-arm, multicenter study to evaluate the efficacy and safety of MK-3475 in patients with ovarian squamous cell carcinoma.

DETAILED DESCRIPTION:
This study includes female patients 18 years of age or older with advanced or recurrent unresectable squamous cell carcinoma of the ovary.

Pembrolizumab will be given for a maximum of 2 years i.e. a total of 35 cycles of pembrolizumab with the q3 week dosing.

ELIGIBILITY:
This study includes female patients 18 years of age or older with advanced or recurrent unresectable squamous cell carcinoma of the ovary. No prior approval (e.g., waiver or exemption) is granted for deviations from the study protocol regarding inclusion criteria.

Inclusion Criteria:

* Participants are eligible to be included in the study only if all of the following criteria apply:

  1. Female participants who are at least 18 years of age on the day of signing informed consent.
  2. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

     1. Not a woman of childbearing potential (WOCBP) as defined OR
     2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
  3. The participant is diagnosed with advanced or recurrent unresectable squamous cell carcinoma of ovary which are histologically confirmed.
  4. The participant provides written informed consent for the trial.
  5. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
  6. Archival tumor tissue sample or newly obtained [core, incisional or excisional] biopsy of a tumor lesion not previously irradiated has been provided. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
  7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
  8. Have adequate organ function as defined in the following. Specimens must be collected within 28 days prior to the start of study intervention.

     * Absolute neutrophil count (ANC) ≥1500/µL
     * Platelets ≥100 000/µL
     * Hemoglobin ≥9.0 g/dL
     * Creatinine ≤1.5 × upper limit of normal (ULN) OR Measured or calculatedb creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN of Creatinine
     * Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
     * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
     * PT - International normalized ratio (INR) < 1.5
     * Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

9.1 Hepatitis B positive subjects

* Participants who are HBsAg positive are eligible if they have received Hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization.
* Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.

9.2 Hepatitis C positive subjects

* Participants with history of Hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening.
* Participants must have completed curative anti-viral therapy at least 4 weeks prior to randomization.

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:

  1. A WOCBP who has a positive serum or urine pregnancy test within 72 hours prior to registration .
  2. TMB-High (TMB score ≥ 10 mut/Mb) by FoundationOne CDx Cancer Genome Profile.
  3. MSI-High by microsatellite instability test or FoundationOne CDx Cancer Genome Profile.
  4. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
  5. Has received prior systemic anti-cancer therapy including investigational agents within 28 days prior to registration.

     Note: There is no limit to the number of chemotherapy treatments prior to the study. Participants must have recovered from all adverse events (AE) due to previous therapies to ≤Grade 1 or baseline. Participants with alopecia and ≤Grade 2 neuropathy may be eligible. Participants with endocrine-related AE Grade ≤2 requiring treatment or hormone replacement may be eligible Note: If the participant had major surgery, the participant must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention.
  6. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
  7. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.

     Note: please refer to Section 5.4.2 for information on COVID-19 vaccines
  8. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.

     Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
  9. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
  10. Known additional malignancy that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
  11. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
  12. Has severe hypersensitivity (≥Grade 3) to MK-3475 and/or any of its excipients.
  13. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
  14. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
  15. Has an active infection requiring systemic therapy.
  16. Has a known history of Human Immunodeficiency Virus (HIV) infection.
  17. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.
  18. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
  19. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
  20. Is pregnant or breast feeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
  21. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 years
  ORR is defined as the proportion of patients with the best overall response to complete response) or partial response (PR) as judged by the blinded independent central review (BICR) according to RECIST 1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  PFS is defined as the time from enrollment to the first recorded point of disease progression (PD) (as assessed by BICR according to RECIST 1.1) or death from any cause, whichever occurs first.For participants that are alive, their survival time will be censored at last disease assessment.
Overall survival (OS) | 2 years
  OS is defined as the time from enrollment to death from any cause.For participants that are alive, their survival time will be censored at the date of last contact.
Duration of response (DOR) | 2 years
  DOR is be defined as the time from the date a response was first documented until the date of disease progression (as assessed by BICR according to RECIST 1.1) or death from any cause, whichever occurs first. For participants that are alive, their survival time will be censored at last disease assessment.
safety and tolerability of MK-3475 therapy | 2 years
  To assess the incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and immune-related adverse events (irAEs), and the proportion of patients discontinuing study treatment due to TEAEs.

OTHER OUTCOMES:
Exploratory objective: molecular biomarkers for MK-3475 therapy for ovarian squamous cell carcinoma. | 2 years
  ORR, PFS, OS, and DOR are assessed in the subgroups divided into high/low XCL1 expression population in tumor tissues, high/low PD-L1 expression population, or high/low tumor infiltration population of CD8 positive lymphocytes.
Tumor shrinkage efficacy is evaluated by investigator according to RECIST1.1 and iRECIST . | 2 years
  ORR is defined as the proportion of patients with the best overall response to CR/iCR or PR/iPR as determined by the investigator based on RECIST1.1 and iRECIST .
  PFS is defined as the time from enrollment to the first recorded point of disease progression (as assessed by investigator according to RECIST1.1 and iRECIST) or death from any cause, whichever occurs first. For participants that are alive, their survival time will be censored at last disease assessment .
  DOR is defined as the time from the date a response was first documented until the date of disease progression (as assessed by investigator according to RECIST1.1 and iRECIST) or death from any cause, whichever occurs first. For participants that are alive, their survival time will be censored at last disease assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Kosuke Yoshihara, Professor, Principal Investigator — Niigata University Medical & Dental Hospital
Locations (1):
- Niigata University Medical & Dental Hosptal, Niigata, Niigata, Japan

IPD SHARING:
Plan to Share IPD: No